CLINICAL TRIAL: NCT06553378
Title: The GOS-Frail (Geriatric Oncology Supportive Care for Frail Older Adults With Cancer) Study
Acronym: GOS-Frail
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: National University of Singapore (Other); National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-3521
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Geriatric Oncology; Supportive Care; Quality of Life
Keywords: Geriatric Oncology; Supportive Care; Quality of Life

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care
- Geriatric Oncology Supportive Clinic (Experimental): Seen at GOSC
  Interventions: Other: Geriatric Oncology Supportive Clinic

INTERVENTIONS:
Other: Geriatric Oncology Supportive Clinic — Subjects in the intervention arm will be seen within four weeks of recruitment. Clinical assessment involves a Comprehensive Geriatric Assessment (CGA) and Supportive Care Assessment conducted by a geriatric-oncologist. Both clinical assessments and targeted interventions are supported by a multi-disciplinary team comprising the geriatrician, geriatric trained nurse, physiotherapist, occupational therapist, speech therapist, pharmacist, dietician, and medical social worker. We will conduct an initial GOSC assessment, with a follow up review during oncology treatment. Subsequently, further GOSC clinic sessions duration of follow up will be determined by the subject's underlying disease, symptom burden and clinical course during treatment.
  Arms: Geriatric Oncology Supportive Clinic

SUMMARY:
Background Cancer is more prevalent in older adults, but most cancer treatment trials have mainly involved young and healthy subjects. Among geriatric syndromes, frailty is a significant risk factor for negative outcomes such as treatment delays, discontinuation, and treatment-related side effects, as well as functional decline and poor survival. Research has shown that geriatric assessment with appropriate intervention can improve these outcomes, although the impact may be influenced by the inclusion of patients receiving palliative-intent treatment. Supportive care focuses on symptom assessment and treatment to enhance treatment tolerance and quality of life. To date, there have been no studies examining the combined benefits of geriatric oncology and supportive care clinics. We conducted a pilot study called Geriatric Oncology Supportive Clinic for Elderly (GOSPEL), which demonstrated an improved quality of life for older adults with curable cancer. Based on these results, we developed an enhanced care model.

Aim The study GOS-Frail aims to assess the effect of an integrated Geriatric Oncology Supportive Clinic on the quality of life of older adults with cancer receiving curative-intent chemotherapy and/or radiotherapy at 1 month.

Methods The GOS-Frail study is a multi-centre, open-label, parallel-arm, randomized controlled trial conducted in the specialist outpatient clinics of two university-affiliated tertiary care hospitals. 154 adults aged 65 and above, diagnosed with solid organ cancer and planned for curative-intent chemotherapy and/or radiotherapy, and with a clinical frailty scale score of 4 and above, will be recruited. Subjects will be randomized to either attend a geriatric oncology supportive clinic or receive frailty education material. Quality of life questionnaires will be administered at baseline, 2 weeks, and 1, 3, 6, and 12 months from treatment initiation.

Hypothesis:

The GOS-Frail study investigates on the role of a synergistic geriatric oncology and supportive model of care in improving quality of life in older adults undergoing curative-intent cancer treatment.

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 65
2. Diagnosis of solid organ cancer
3. Plan for curative-intent chemotherapy and/or radiotherapy
4. Clinical Frailty Scale (CFS) score ≥ 4,

Exclusion criteria: Evaluation by Geriatric or Palliative Medicine in the previous 6 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
EuroQoL-5 Dimension (EQ5D-5L) | 1 month
  EuroQoL-5 Dimension (EQ5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Wen Yang Goh, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No